CLINICAL TRIAL: NCT07027813
Title: Feasibility and Efficacy of Ambulance-Based m-Health for Pediatric Emergencies in Low Resource Settings (FEAMER) Trial
Brief Title: Feasibility and Efficacy of Ambulance-Based m-Health for Pediatric Emergencies (FEAMER) Trial
Acronym: FEAMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-08023879; 4R33HD103049-03 (NIH)
Record Dates: First submitted 2025-06-16; First posted 2025-06-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Emergencies; mHealth; Child Health; Critical Illness
Keywords: Emergency Medical Services; Ambulance; Telemedicine
MeSH Terms: conditions — Emergencies; Critical Illness | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Active Comparator): Patients who are being transported through ambulance but do not receive telemedicine.
  Interventions: Other: Control
- Intervention Group (Experimental): Patients who are transported through ambulance and receive telemedicine support via physicians using mHealth.
  Interventions: Other: Telemedicine
- Telemedicine Physicians (TMPs) (No Intervention): Telemedicine physicians will be providing teleconsultation in the intervention arm for the treatment of pediatric patients during ambulance transport.
- Emergency Medical Technicians (EMTs) (No Intervention): EMTs are trained in both control and intervention settings. The delivery of intervention will depend on the ambulance that they will be operating in during the transport.

INTERVENTIONS:
Other: Telemedicine — Provision of Telemedicine support to pediatric patients during ambulance transport.
  Other Names: mHealth
  Arms: Intervention Group
Other: Control — Provision of ambulance transport without any telemedicine support.
  Other Names: Simple Ambulance transport
  Arms: Control Group

SUMMARY:
Investigators hypothesize that in a low-resource setting, linking ambulances that transport acutely ill children to a remote pediatric emergency physician using a simple audio-video device will improve the quality of these children's medical decisions and health outcomes. For this purpose, the investigators will conduct a study in Karachi, Pakistan, where they will collect medical data for ill children at the time of ambulance pickup, hospital drop-off, and during hospital triage. During transport, one group will receive a telemedicine call from a trained physician, while the other group will receive basic paramedic treatment. The investigators will then compare both groups.

DETAILED DESCRIPTION:
Background:

Almost half of all 6.2 million deaths in children worldwide are caused by acute illnesses such as pneumonia, diarrhea, and injuries, and occur disproportionately in low- and middle-income countries (LMICs). These acute illnesses are mostly treatable if diagnosed and managed in a timely fashion. According to estimates, about half of these children can be saved through better emergency care.

Emergency medical care at the scene and during transportation is, therefore, critical to improving health outcomes. The "Chain of Survival" for cardiac arrest, the "Golden hour" of trauma, and the "FAST" program for stroke rely heavily on high-quality Emergency Medical Systems (EMS). For many emergency conditions, triage and care decisions during transportation play a critical role in the eventual outcome. EMS staff well-trained in pediatric acute/emergency care are scarce, even in high-income countries, and essentially non-existent in LMICs.

There is a critical need - globally, but particularly in LMICs - to address this expertise gap during the most critical time period while a child is transported to a fixed emergency care facility. Such solutions can contribute to potentially saving thousands of children every year.

Formal EMS systems consist of a universal access number (such as 911) that connects the community to ambulances equipped with the necessary supplies, protocols, and, most importantly, trained healthcare providers through specialized call centers. In low-resource settings, the contribution of effective transportation to health outcomes becomes far more significant. Studies show that the lack of EMS contributed to two-thirds of all trauma deaths, 52% of maternal and perinatal deaths, and 20% of newborn deaths in LMICs. Mobile health technology available today has the potential to bridge the expertise gap in prehospital settings rapidly. While there is a sound theoretical basis for such intervention, there is no evidence on the use of ambulance-based teleconsultation (ABT) for children.

Pakistan, the setting of this study, ranks third in the number of deaths among children. On average, every twelfth child who dies worldwide is a Pakistani child. Unpublished data from Karachi, Pakistan, shows a very high acuity level amongst children transported by ambulances. The only modern ambulance service and our partner in this project, Sindh Integrated Emergency & Health Services (SIEHS), transported 36,501 children between Jan 1, 2018, and Dec 31, 2019. Of these, 12,200 (33%) were triaged as serious or life-threatening emergencies using the globally accepted standard called the Medical Priority Dispatch System.

The current process of care of the critically ill child: Currently, when a family calls the SIEHS Universal Access Number (1021), the call taker/dispatcher team in the Command-and-Control Center (CCC) asks a set of standard questions to determine the patient's location and estimate the potential severity of their condition. The dispatcher then locates the nearest ambulance and passes on the location information and severity code to the ambulance crew. Upon arrival at the scene, EMTs provide emergency care in accordance with established clinical protocols until they reach the destination hospital. The ambulance staff "signs out" patients to the hospital staff, sharing their history and any treatment provided.

Through this study, the investigators aim to test the efficacy of ABT by measuring a change in the outcome measure of PEWS for acutely ill children from the scene of injury/illness to the pediatric emergency department (PED) through a cluster-randomized trial.

Study Procedures:

We will randomly assign 60 ambulances to control and ABT intervention groups (30 each) using a stratified random sampling design. We will assign 30 ambulances, five from each of the six administrative zones of SIEHS, to receive the ABT setup. We will compare changes in PEWS as noted by EMTs at the scene of illness/injury and the PEWS noted by triage nurses in the emergency department between the ABT and control groups.

Sample Size:

For this study, a total of 600 children will be enrolled. All EMTs at the SIEHS (~272 currently) and all telemedicine physicians at CLF(24 currently) will be included in delivering the intervention. For pediatric patients, we based our sample size calculation on the ability to detect a clinically significant difference as captured by a medium to large effect size (0.6-0.8). We estimate that a total sample size of 600 patients will be required for the study (300 in each arm) to detect a medium to significant difference with a standard deviation of 2.0-3.0, a power of 80%, and a significance level of 0.05 (two-sided).

Recruitment:

Patients transported by the intervention ambulances will be enrolled in the intervention arm, while those transported by the control ambulances will be in the control arm. The distribution of patients to these ambulances is random based on the location of the patient and the ambulance at the time of the emergency call. Upon arrival, a trained EMT will approach the parents/guardians, make an initial assessment for eligibility, explain the study intervention, and recruit them to the interventional or control group.

Parents will be consented to by the EMTs. EMTs who will obtain consent will receive training on effective communication and the appropriate approach to obtaining consent from parents for research studies. Based on our preliminary qualitative study findings, we will obtain written consent followed by an opt-out strategy.

The right to withdraw from the study will be respected. Parents can withdraw from the study by contacting the research through a telephone contact number they will receive during the consent process. Additionally, the research team will contact all participants after 72 hours and offer them another opportunity to withdraw from the study. If participants do not withdraw during the call by the study team or by the data lock date, their data will be de-identified and included in the analysis.

Equipment Installation:

The SIEHS, CLF, and AKU (Aga Khan University) teams (in coordination with our human-factor engineering consultant, PD) are responsible for the selection and installation of equipment. The study investigators have equipped ambulances in the intervention arm for real-time, bi-directional, audio-video communication, allowing virtual interactions between EMTs, patients, caretakers, and TMPs; 1- An IP phone with a 4G router supports the communication and connection with the TMPs, 2- To ensure hand-free interaction with the patients, all EMTs wear a headset to communicate with the TMPs, 3- The 360 rotation camera has been installed to allow live video transmission to TMP. The video stream has been integrated into the pre-existing telemedicine platform at CLF through their proprietary software. 4- A tablet with a Qualtrics form has been installed in the ambulance for recording consent and PEWS data. 5- A 4G internet device with a router is present in all ambulances to allow constant signals.

Investigators have utilized existing data privacy standards at CLF to ensure password-protected login, role-based access control, secure Hypertext Transfer Protocol (HTTP) encryption, and data transfer through a virtual private network (VPN). All installed equipment undergoes a quality check and is certified in accordance with local standards before use. If device troubleshooting is required, technical assistance is provided in person or remotely, as needed. Equipment evaluation is collected in the SIEHS equipment checklist, and the following variables are assessed: phone, camera, and tablet.

Data Collection:

We will use the Modified Brighton PEWS as the outcome indicator to test the effectiveness of ABT on patient outcomes. The standard PEWS table has been added to the current clinical form of SIEHS and triage form at CLF EDs. EMTs will obtain consent, calculate the PEWS score, communicate the initial PEWS scores to the SIEHS command and control center, and enter them in the Qualtrics form provided by the WCM. At the time of drop off, the second set of PEWS will be entered on Qualtrics by the EMT, and the child will be handed over to the hospital. Every morning, the SMRS data coordinator will email an Excel spreadsheet of all cases transferred by SMRS to CLF hospitals. Simultaneously, CLF will calculate the triage PEWS and share it with the study coordinator at WCM. The difference in PEWS score (primary outcome), as measured by EMTs from initial evaluation, drop-off evaluation, and ED triage, will be calculated and compared between patients receiving regular care and those receiving ABT consultation.

ELIGIBILITY:
CHILDREN

Inclusion criteria:

* Age 0-14 years
* Children transported by an SIEHS ambulance with a transport time of ≥20 minutes
* Children presenting to the ChildLife Emergency Department with a parent/ guardian present in the ambulance to consent
* Children classified as "Charlie, Delta, Echo" on the Medical Priority Dispatch System

Exclusion Criteria:

• Children transported without an adult parent or guardian

EMERGENCY MEDICAL TECHNICIANS (EMTs)

Inclusion Criteria:

• EMTs currently employed by the SIEHS EMS service.

Exclusion Criteria:

• EMTs who refuse to participate or consent to the study.

TELEMEDICINE PHYSICIANS (TMPs)

Inclusion Criteria:

• TMPs currently employed by the CLF Telemedicine services.

Exclusion Criteria:

• TMPs who refuse to participate or consent to the study.

Ages: 1 Minute to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Early Warning Signs (PEWS) Score | At the ambulance pick up and hospital drop off (>20 minutes)
  PEWS Score is "0" for a normal patient, and ranges between "1-9" depending upon severity of illness i.e., higher PEWS scores referring to higher severity of illness. Modified Brighton PEWS used in our study accounts for Respiratory rate, Heart Rate, and Appearance.
Pediatric Early Warning Signs (PEWS) Score at the ambulance drop off | At the ambulance drop off (>20 minutes)
  PEWS Score is "0" for a normal patient, and ranges between "1-9" depending upon severity of illness i.e., higher PEWS scores referring to higher severity of illness. Modified Brighton PEWS used in our study accounts for Respiratory rate, Heart Rate, and Appearance.

SECONDARY OUTCOMES:
Percent of completed Telemedicine Calls | During ambulance ride (>20 minutes)
Satisfaction of Emergency Medical Technicians and Telemedicine Physicians as measured by the System Usability Survey | 1 month after the end of trial i.e., completion of study
  10 questions with a likert scale ranging from 1-5, with a higher score indicating better perceived usability.
Outcome at end of Emergency Department (ED) Visit | On arrival to the ED triage
  ED mortality
72 hour outcome after the Emergency Department (ED) Visit | Within 72 hours of reaching the ED
  72 hour mortality after admission to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Junaid Razzak, MD,PhD,FACEP, Principal Investigator — Weill Cornell School of Medicine, NY
Locations (3):
- Pakistan (3):
  - Aga Khan University Hospital, Karachi, Sindh
  - ChildLife Foundation, Karachi, Sindh
  - Sindh Integrated Emergency and Health Services (SIEHS), Karachi, Sindh

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual Patient Data (IPD) that underlies results will be submitted in a report format to NIH and published in well-reputed journals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available at the end of trial completion when the findings are submitted to Eunice Kennedy Shriver National Institute of Child Health and Human Development in the form of a detailed report.
Access Criteria: The data will be accessible upon request to the Principal investigator for researchers who intend to learn, adapt, or replicate from our trial findings.

REFERENCES:
- [Background] Levels and trends in child mortality 2015. New York: 1. United Nations Children's Fund (UNICEF). 2015.
- [Background] Committing to Child Survival: A Promise Renewed: Progress Report 2014. New York: 1. United Nations Children's Fund (UNICEF). 2014.
- [Background] Ahrens T. Extravascular lung water. Concepts in clinical application. Crit Care Nurs Clin North Am. 1989 Dec;1(4):681-8. PMID 2627321
- [Background] GBD Results Tool, GHDx, IHME. 2019; http://ghdx.healthdata.org/gbd-results-tool. Accessed November 1, 2019
- [Background] International Statistical Classification of Diseases and Related Health Problems (ICD-11). 25 May 20192019;Newsroom.
- [Background] Thaddeus S, Maine D. Too far to walk: maternal mortality in context. Soc Sci Med. 1994 Apr;38(8):1091-110. doi: 10.1016/0277-9536(94)90226-7. PMID 8042057
- [Background] Hsia RY, Thind A, Zakariah A, Hicks ER, Mock C. Prehospital and Emergency Care: Updates from the Disease Control Priorities, Version 3. World J Surg. 2015 Sep;39(9):2161-7. doi: 10.1007/s00268-015-2997-5. PMID 25847225
- [Background] Mock CN, Jurkovich GJ, nii-Amon-Kotei D, Arreola-Risa C, Maier RV. Trauma mortality patterns in three nations at different economic levels: implications for global trauma system development. J Trauma. 1998 May;44(5):804-12; discussion 812-4. doi: 10.1097/00005373-199805000-00011. PMID 9603081
- [Background] Krug EG, Sharma GK, Lozano R. The global burden of injuries. Am J Public Health. 2000 Apr;90(4):523-6. doi: 10.2105/ajph.90.4.523. PMID 10754963
- [Background] Mawani M, Kadir MM, Azam I, Mehmood A, McNally B, Stevens K, Nuruddin R, Ishaq M, Razzak JA. Epidemiology and outcomes of out-of-hospital cardiac arrest in a developing country-a multicenter cohort study. BMC Emerg Med. 2016 Jul 28;16(1):28. doi: 10.1186/s12873-016-0093-2. PMID 27465304
- [Background] Merali HS, Lipsitz S, Hevelone N, Gawande AA, Lashoher A, Agrawal P, Spector J. Audit-identified avoidable factors in maternal and perinatal deaths in low resource settings: a systematic review. BMC Pregnancy Childbirth. 2014 Aug 16;14:280. doi: 10.1186/1471-2393-14-280. PMID 25129069
- [Background] Waiswa P, Kallander K, Peterson S, Tomson G, Pariyo GW. Using the three delays model to understand why newborn babies die in eastern Uganda. Trop Med Int Health. 2010 Aug;15(8):964-72. doi: 10.1111/j.1365-3156.2010.02557.x. PMID 20636527
- [Background] Alkire BC, Raykar NP, Shrime MG, Weiser TG, Bickler SW, Rose JA, Nutt CT, Greenberg SL, Kotagal M, Riesel JN, Esquivel M, Uribe-Leitz T, Molina G, Roy N, Meara JG, Farmer PE. Global access to surgical care: a modelling study. Lancet Glob Health. 2015 Jun;3(6):e316-23. doi: 10.1016/S2214-109X(15)70115-4. Epub 2015 Apr 27. PMID 25926087
- [Background] Krnjevic K, Morris ME. An excitatory action of substance P on cuneate neurones. Can J Physiol Pharmacol. 1974 Jun;52(3):736-44. doi: 10.1139/y74-094. No abstract available. PMID 4850541
- [Background] Gausche-Hill M, Ely M, Schmuhl P, Telford R, Remick KE, Edgerton EA, Olson LM. A national assessment of pediatric readiness of emergency departments. JAMA Pediatr. 2015 Jun;169(6):527-34. doi: 10.1001/jamapediatrics.2015.138. PMID 25867088
- [Background] Houston R, Pearson GA. Ambulance provision for children: a UK national survey. Emerg Med J. 2010 Aug;27(8):631-6. doi: 10.1136/emj.2009.088880. Epub 2010 Jun 1. PMID 20515914
- [Background] Patterson PD, Baxley EG, Probst JC, Hussey JR, Moore CG. Medically unnecessary emergency medical services (EMS) transports among children ages 0 to 17 years. Matern Child Health J. 2006 Nov;10(6):527-36. doi: 10.1007/s10995-006-0127-6. Epub 2006 Jul 1. PMID 16816999
- [Background] Seidel, J. S., & Henderson, D. P. (Eds.). (1991). Emergency medical services for children: a report to the nation. National Center for Education in Maternal and Child Health.
- [Background] Kironji AG, Hodkinson P, de Ramirez SS, Anest T, Wallis L, Razzak J, Jenson A, Hansoti B. Identifying barriers for out of hospital emergency care in low and low-middle income countries: a systematic review. BMC Health Serv Res. 2018 Apr 19;18(1):291. doi: 10.1186/s12913-018-3091-0. PMID 29673360
- [Background] Sriram V, Gururaj G, Razzak JA, Naseer R, Hyder AA. Comparative analysis of three prehospital emergency medical services organizations in India and Pakistan. Public Health. 2016 Aug;137:169-75. doi: 10.1016/j.puhe.2016.02.022. Epub 2016 Apr 12. PMID 27080583
- [Background] Zafar W, Siddiqui E, Ejaz K, Shehzad MU, Khan UR, Jamali S, Razzak JA. Health care personnel and workplace violence in the emergency departments of a volatile metropolis: results from Karachi, Pakistan. J Emerg Med. 2013 Nov;45(5):761-72. doi: 10.1016/j.jemermed.2013.04.049. Epub 2013 Sep 4. PMID 24011477
- [Background] Jewkes F. Prehospital emergency care for children. Arch Dis Child. 2001 Feb;84(2):103-5. doi: 10.1136/adc.84.2.103. No abstract available. PMID 11159280
- [Background] Rortgen D, Bergrath S, Rossaint R, Beckers SK, Fischermann H, Na IS, Peters D, Fitzner C, Skorning M. Comparison of physician staffed emergency teams with paramedic teams assisted by telemedicine--a randomized, controlled simulation study. Resuscitation. 2013 Jan;84(1):85-92. doi: 10.1016/j.resuscitation.2012.06.012. Epub 2012 Jun 30. PMID 22750663
- [Background] Brokmann JC, Conrad C, Rossaint R, Bergrath S, Beckers SK, Tamm M, Czaplik M, Hirsch F. Treatment of Acute Coronary Syndrome by Telemedically Supported Paramedics Compared With Physician-Based Treatment: A Prospective, Interventional, Multicenter Trial. J Med Internet Res. 2016 Dec 1;18(12):e314. doi: 10.2196/jmir.6358. PMID 27908843
- [Background] Lippman JM, Smith SN, McMurry TL, Sutton ZG, Gunnell BS, Cote J, Perina DG, Cattell-Gordon DC, Rheuban KS, Solenski NJ, Worrall BB, Southerland AM. Mobile Telestroke During Ambulance Transport Is Feasible in a Rural EMS Setting: The iTREAT Study. Telemed J E Health. 2016 Jun;22(6):507-13. doi: 10.1089/tmj.2015.0155. Epub 2015 Nov 24. PMID 26600433
- [Background] Skorning M, Bergrath S, Rortgen D, Beckers SK, Brokmann JC, Gillmann B, Herding J, Protogerakis M, Fitzner C, Rossaint R; Med-on-@ix-Working Group. Teleconsultation in pre-hospital emergency medical services: real-time telemedical support in a prospective controlled simulation study. Resuscitation. 2012 May;83(5):626-32. doi: 10.1016/j.resuscitation.2011.10.029. Epub 2011 Nov 22. PMID 22115932
- [Background] Lenssen N, Krockauer A, Beckers SK, Rossaint R, Hirsch F, Brokmann JC, Bergrath S. Quality of analgesia in physician-operated telemedical prehospital emergency care is comparable to physician-based prehospital care - a retrospective longitudinal study. Sci Rep. 2017 May 8;7(1):1536. doi: 10.1038/s41598-017-01437-5. PMID 28484212
- [Background] Brokmann JC, Rossaint R, Muller M, Fitzner C, Villa L, Beckers SK, Bergrath S. Blood pressure management and guideline adherence in hypertensive emergencies and urgencies: A comparison between telemedically supported and conventional out-of-hospital care. J Clin Hypertens (Greenwich). 2017 Jul;19(7):704-712. doi: 10.1111/jch.13026. Epub 2017 May 30. PMID 28560799
- [Background] Institute Of Medicine. IOM report: the future of emergency care in the United States health system. Acad Emerg Med. 2006 Oct;13(10):1081-5. doi: 10.1197/j.aem.2006.07.011. No abstract available. PMID 17015421
- [Background] Price CI, Shaw L, Dodd P, Exley C, Flynn D, Francis R, Islam S, Javanbakht M, Lakey R, Lally J, McClelland G, McMeekin P, Rodgers H, Snooks H, Sutcliffe L, Tyrell P, Vale L, Watkins A, Ford GA. Paramedic Acute Stroke Treatment Assessment (PASTA): study protocol for a randomised controlled trial. Trials. 2019 Feb 12;20(1):121. doi: 10.1186/s13063-018-3144-z. PMID 30755249
- [Background] Robinson MJ, Taylor J, Brett SJ, Nolan JP, Thomas M, Reeves BC, Rogers CA, Voss S, Clout M, Benger JR; AIRWAYS-2 study team. Design and implementation of a large and complex trial in emergency medical services. Trials. 2019 Feb 8;20(1):108. doi: 10.1186/s13063-019-3203-0. PMID 30736841
- [Background] Dishaw, M. T., & Strong, D. M. (1999). Extending the technology acceptance model with task- technology fit constructs. Information & management, 36(1), 9-21.
- [Background] Zakria M, Muhammad F. Forecasting the population of Pakistan using ARIMA models. Pakistan Journal of Agricultural Sciences. 2009;46(3):214-223.
- [Background] Kazmi JH, Zubair S. Estimation of vehicle damage cost involved in road traffic accidents in Karachi, Pakistan: a geospatial perspective. Procedia engineering. 2014;77:70-78.
- [Background] Sriram VM, Naseer R, Hyder AA. Provision of prehospital emergency medical services in Punjab, Pakistan: Case study of a public sector provider. Surgery. 2017 Dec;162(6S):S12-S23. doi: 10.1016/j.surg.2017.02.015. Epub 2017 May 15. PMID 28522129
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Addissie A, Davey G, Newport MJ, Addissie T, MacGregor H, Feleke Y, Farsides B. A mixed-methods study on perceptions towards use of Rapid Ethical Assessment to improve informed consent processes for health research in a low-income setting. BMC Med Ethics. 2014 May 2;15:35. doi: 10.1186/1472-6939-15-35. PMID 24885049
- [Background] Mwaka E, Nakigudde J, Ali J, Ochieng J, Hallez K, Tweheyo R, Labrique A, Gibson DG, Rutebemberwa E, Pariyo G. Consent for mobile phone surveys of non-communicable disease risk factors in low-resource settings: an exploratory qualitative study in Uganda. Mhealth. 2019 Aug 19;5:26. doi: 10.21037/mhealth.2019.07.05. eCollection 2019. PMID 31559271
- [Background] Deja E, Peters MJ, Khan I, Mouncey PR, Agbeko R, Fenn B, Watkins J, Ramnarayan P, Tibby SM, Thorburn K, Tume LN, Rowan KM, Woolfall K. Establishing and augmenting views on the acceptability of a paediatric critical care randomised controlled trial (the FEVER trial): a mixed methods study. BMJ Open. 2021 Mar 10;11(3):e041952. doi: 10.1136/bmjopen-2020-041952. PMID 33692177
- [Background] Weijer C, Grimshaw JM, Eccles MP, McRae AD, White A, Brehaut JC, Taljaard M; Ottawa Ethics of Cluster Randomized Trials Consensus Group. The Ottawa Statement on the Ethical Design and Conduct of Cluster Randomized Trials. PLoS Med. 2012;9(11):e1001346. doi: 10.1371/journal.pmed.1001346. Epub 2012 Nov 20. PMID 23185138
- [Background] Woolfall K, Frith L, Dawson A, Gamble C, Lyttle MD; CONNECT advisory group; Young B. Fifteen-minute consultation: an evidence-based approach to research without prior consent (deferred consent) in neonatal and paediatric critical care trials. Arch Dis Child Educ Pract Ed. 2016 Feb;101(1):49-53. doi: 10.1136/archdischild-2015-309245. Epub 2015 Oct 13. No abstract available. PMID 26464416
- [Background] Offerman SR, Nishijima DK, Ballard DW, Chetipally UK, Vinson DR, Holmes JF. The use of delayed telephone informed consent for observational emergency medicine research is ethical and effective. Acad Emerg Med. 2013 Apr;20(4):403-7. doi: 10.1111/acem.12117. PMID 23701349
- [Background] Babchuk WA. Glaser or Strauss? Grounded theory and adult education. Paper presented at: Proceedings of the 15th Annual Midwest Research-to-Practice Conference in Adult, Continuing, and Community Education1996.
- See also: Sindh Rescue and Medical Services launched at the Sindh Secretariat: Aman Foundation — https://www.siehs.org/
- See also: ChildLife Foundation (CLF) — http://childlifefoundation.org/